CLINICAL TRIAL: NCT00006272
Title: Study of Energy Expenditure in Infants With Ventricular Septal Defects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Indiana University School of Medicine (Other)
Other Study IDs: NCRR-M01RR00750-9045; IU-9607-08; IU-9511-16
Record Dates: First submitted 2000-09-11; First posted 2000-09-12 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Heart Septal Defects, Ventricular
Keywords: cardiovascular and respiratory diseases; heart defects; rare disease
MeSH Terms: conditions — Heart Septal Defects, Ventricular; Respiratory Tract Diseases; Rare Diseases

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
OBJECTIVES:

I. Compare the total daily energy expenditure in infants with ventricular septal defects vs healthy control infants.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Height, weight, and vital signs (including oxygen saturation by pulse oximetry) are measured on Day 1. Resting energy expenditure, oxygen consumption (VO2), carbon dioxide production (VCO2), and resting respiratory exchange quotient (RQ) are measured using open circuit respiratory calorimetry on Day 1. Patients undergo assessment of total daily energy expenditure using the doubly labeled water method comprised of oral deuterium and oral oxygen O 18 with the next scheduled feeding on Day 1. Urine samples are collected prior to isotope administration, then serially for approximately 12 hours after isotope administration on Day 1, and then daily on Days 2-7. These samples are analyzed by mass spectrometry. On Day 1, patients also undergo echocardiogram to confirm size of defect and measure the degree of pulmonary/systemic blood flow ratio and pulmonary artery pressures.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Infants with moderate to large ventricular septal defect (VSD) by most recent echocardiogram who meet the following conditions: no other concurrent heart or lung disease; no chromosomal defects or congenital anomalies

OR

Healthy control infants without VSD who meet the following conditions: clinically well; no heart disease; no chromosomal defects or congenital anomalies

--Prior/Concurrent Therapy--

Surgery: VSD infants -- No prior cardiac surgery or palliative procedures; VSD and control infants -- Greater than 6 weeks since other prior surgery

Other: VSD and control infants: Greater than 6 weeks since prior hospitalization

Ages: 3 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20
Dates: Start 1994-08

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A. Leitch, Study Chair — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States